CLINICAL TRIAL: NCT06116097
Title: The Effect of Nutrition Education Sessions on Energy Availability, Body Composition, Eating Attitude and Sports Nutrition Knowledge in Young Female Endurance Athletes
Brief Title: Effect of Nutrition Education on Energy Availability, Body Composition, Eating Attitude and Sports Nutrition Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Cansu Tektunalı Akman, Mrs., Medipol University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: E.8234/196
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Relative Energy Deficiency in Sport
MeSH Terms: conditions — Relative Energy Deficiency in Sport | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A total of 83 adolescent female elite athletes from 3 different sport clubs (football n=34, basketball n=16 and volleyball n=33) between 15 and 18 years(mean 17.2 ± 2.0) were included in the study.They were divided into either the intervention or the control groupby simple randomization. Fortyfem participants took 6 physical nutrition education lectures and the other group (n=38) didn't have any nutrition education. All of them filled the LEAF-Q (Low energy availability in athletes questionnaire),EAT-26(Eating Attitude Test)and SNKQ (Sports Nutrition Knowledge Questionnaire).Energy and nutrient intakes were assessed based on 3-day food records. Activity logs were analysed to measure exercise energy expenditure. All of the tests have been repeated after 6 months. Nutrition education was comprised of 6 physical 60 minutes sessions given every week in a school class. Each session was consisted of a different subject. Participants got written information as a printed booklet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition education intervention group (Experimental): Nutrition education was comprimised of 6 physical face to face 60 minutes sessions which was given every week in a school class. Each session was consisted of a different subject including energy metabolism in sport, energy balance, nutrition before and after training, low energy availability, macro and micronutrients, hydration and supplements. Participants also got written information as a printed booklet in order to be able to take notes under sessions and review after the sessions.
  Interventions: Behavioral: Nutrition education
- Control group (No Intervention): Control group has not taken any nutrition education but has been filled all of the questionnaires, acitivity logs and food diaries.

INTERVENTIONS:
Behavioral: Nutrition education — Fifty participants took 6 physical nutrition education lectures and the other group (n=33) didn't have any nutrition education. Nutrition education was comprimised of 6 physical face to face 60 minutes sessions which was given every week in a school class. Each session was consisted of a different subject including energy metabolism in sport, energy balance, nutrition before and after training, low energy availability, macro and micronutrients, hydration and supplements. Participants also got written information as a printed booklet in order to be able to take notes under sessions and review after the sessions.
  Arms: Nutrition education intervention group

SUMMARY:
This study investigates the effects of a series of nutrition education sessions conducted by a registered dietitian on energy availability, various anthropometric measurements, eating attitudes, and sports nutrition knowledge in young female endurance athletes aged 15-18 years (football, basketball, volleyball) who engage in training for more than 10 hours per week (n=83).

DETAILED DESCRIPTION:
Participants were randomly divided into two groups with 45 individuals receiving six physical nutrition education lectures, and the remaining 38 participants receiving no nutrition education. Participants completed the The low energy availability in females questionnaire (LEAF-Q), Eating Attitude Test (EAT-26) and Sports Nutrition Knowledge Questionnaire (SNKQ). Energy and nutrient intakes were evaluated thorough 3-day food records, while exercise energy expenditure was assessed using 3-day activity logs. All of the questionnaires were repeated after a 6-months period.

At baseline, the prevalence of LEA among athletes was determined to be 63.8%. In the intervention group, energy availability (EA) and SNKQ scores increased, and LEAF-Q scores decreased significantly (p < 0.05). However, there was no significant change in EAT-26 scores between the two groups. Energy intake, weight, fat free mass and resting metabolic rate has been increased significantly in the intervention group (p < 0,05). These findings suggest that nutrition education proves beneficial in enhancing dietary intake, positively influencing body composition and improving nutrition knowledge, ultimately contributing to increased energy availability in female athletes over the short term.

ELIGIBILITY:
Inclusion Criteria:

Non-contraceptive using Competitive female endurance athletes 14-18 years of age training minimum 6 hours a week not taking a break from sports for more than 3 months due to injury

Exclusion Criteria:

Pregnancy or planned pregnancy chronic diseases (e.g. diabetes, crohn's disease, thyroid dysfunction) Use of any medication that may disturb hormonal balance

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Energy Availability | 6 months
  Energy availability (EA) is described as the amount of energy left over and available for proper organism functions after the energy used for exercise is subtracted from the calories taken in the diet, by American College of Sports Medicine. It is shown that the young athletes often fail to follow the recommended dietary guidelines for their sport and activity level. Therefore that poses risk for low energy availability (LEA) EA below 30 kcal/kg FFM was considered to be low EA, EA between 30-45 kcal/kg was considered to be reduced and EA>45 kcal/kg was considered to be optimal.
Low Energy Availability Questionnaire (LEAF-Q) | 6 months
  The 25-item LEAF-Q was used to assess the risk of LEA. The LEAF-Q has been validated in female athletes aged 18-39 training ≥5 times/week, with findings producing an acceptable sensitivity (78%) and specificity (90%) to classify current energy availability[28]. Consistent with the original validation study players completed a paper version of the LEAF-Q to ensure validity and reliability were maintained. Scoring was based on the original validation study, with those who scored ≤7 being classified as 'not at risk' of LEA, and those who scored ≥8 being classified as 'at risk' of LEA[28].

SECONDARY OUTCOMES:
Sports nutrition knowledge questionnaire (SNKQ) | 6 months
  Players completed the 88-item Sports Nutrition Knowledge Questionnaire (SNKQ) at pre and post intervention.The SNKQ has been assessed for validity (content and construct) and reliability (test-retest), with findings indicating a high construct validity and good test-retest concordance and therefore suitability to be used to determine sports nutrition knowledge. The SNKQ consists of five sub-sections (general nutrition concepts, fluid, recovery, weight control and supplements). One point was awarded for each correct answer, and an 'unsure' or incorrect response received zero points. The scores for each subsection and total score were calculated based on the number of questions answered correctly with a maximum total score of 83.
Eating Atittude Test (EAT-26) | 6 months
  EAT-26 has been used to assess eating disorder risks in many populations, including athletes. As recommended by the developers of the EAT-26 tool, scores of 20 or above on the EAT-26 assessment indicated eating disorder behaviors. Scores falling below 20 were assessed as low risk for eating disorder behaviors
Dietary intake | 6 months
  The mean daily intake of energy, macronutrients and some of the micronutrients over the three days (two weekdays, one weekend) was calculated. Participants used household measures to estimate intake. Dietary intake data was entered into BEBIS 6.1 nutrition analysis program. (Beslenme Bilgi sistemi, Turkey) Daily energy, protein, carbohydrate, fat and fiber intake was compared with the values reported in the current nutrition guidelines.
Exercise Energy Expenditure | 6 months
  Exercise energy expenditure (EEE) has been calculated according to the 3-day activity logs in the beginning of the season. Activity logs (including activity, exercise duration and rest periods) for resistance and any non-club based activities under 3 days were completed and assigned a Metabolic Equivalent (MET) value from the compendium of physical activities
Fat-free mass | 6 months
  at-free mass (FFM) is the primary determinant of TEE in all age groups.
Body Mass Index (BMI) | 6 months
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters.Low BMI was defined as BMI <18.5 kg/m2 as recommended when screening athletes for risk of LEA.
Basal metabolic rate (BMR) | 6 months
  he amount of energy expended while at rest in a neutrally temperate environment, and in a post-absorptive state (meaning that the digestive system is inactive, which requires about 12 hours of fasting)
Fat mass | 6 months
  Body fat can be predictor for eating disorder risk status.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu T Akman, MS, Principal Investigator — Medipol University
Locations (1):
- Baltalimanı Research and Training Hospital, Istanbul, Sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No